CLINICAL TRIAL: NCT05513313
Title: Prospective Assessment of Myocarditis After Replication-Deficient Smallpox Immunization
Brief Title: Assessment of Myocarditis After Replication-Deficient Smallpox Immunization
Acronym: PAMARDSI
Status: Not yet recruiting | Type: Observational
Sponsor: Womack Army Medical Center (U.S. Federal Agency)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency); C.R.Darnall Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laurie Housel, MSN, FNP-C, Womack Army Medical Center
Other Study IDs: PAMARDSI
Record Dates: First submitted 2022-05-02; First posted 2022-08-24 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Myopericarditis; Small Pox
Keywords: Small pox vaccine; ACAM2000™; Dryvax®
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Jynneos vaccine with out other vaccines: Allocated to Jynneos without any need for additional indicated/required vaccines intervention. JYNNEOS (Smallpox and Monkeypox Vaccine, Live, Nonreplicating) suspension for subcutaneous injection. Administer two doses (0.5 mL each) 4 weeks apart. Each dose (0.5 mL) is supplied in a singledose vial.
  Interventions: Biological: JYNNEOS
- Jynneos vaccine with other vaccines at dose 1: Allocated to Jynneos with concomitant vaccines given at time of first dose of Jynneos intervention.
  Interventions: Biological: JYNNEOS
- Jynneos vaccine with other vaccines at dose 2: Allocated to Jynneos with concomitant vaccines given at time of second dose of Jynneos.
  Interventions: Biological: JYNNEOS

INTERVENTIONS:
Biological: JYNNEOS — smallpox vaccine

SUMMARY:
This is a prospective observational phase IV study of a novel, replication-deficient smallpox vaccine that has been recently been approved by FDA. The purpose of this study is to determine if there are any abnormalities detected by electrocardiographic testing and/or blood tests within 35 days of receiving the second dose of smallpox vaccine either alone or co-administered with other vaccines that may/may not be suggestive of myopericarditis.

DETAILED DESCRIPTION:
Receipt of the novel smallpox vaccine JYNNEOS® is a requirement for study participation. Prior to enrollment, potential participants will complete a routine adult immunization screening questionnaire (standard of care) and be reviewed by study team for eligibility prior to enrollment.

The entry questionnaires and copy of medical treatment facility (MTF) records and/or Immunization Tracking System documentation will provide baseline demographic and past medical history with specific attention paid to prior immunization history, past medical history of known atopy, HIV disease, coronary artery disease or myocardial infarction, diabetes, carotid artery disease, stroke, or other cardiac disease risk factors such as hyperlipidemia, smoking, hypertension, obesity, etc. All medications being taken prior to enrollment and throughout the study will be documented. The symptom diary/survey will serve as the vehicle to identify symptom and medication changes during study participation. Subjects will use the Defense and Veterans rating scale to rate their pain. The smallpox entry questionnaire, symptom diary and medication log are study-related. A routine screening immunization questionnaire will be completed and the screening form must not have any contraindication identified for the JYNNEOS® vaccine for consideration of enrollment (standard of care). Laboratory tests and ECGs are not standard of care for receiving smallpox vaccination, but are study-related. Participants who develop new onset cardiac symptoms or other symptoms suggestive of possible cardiac involvement which might meet the CDC/DoD case definition of suspect, probable or confirmed myopericarditis, will be referred to Defense Health Agency-Immunization Healthcare Division (DHA-IHD) clinical team as well as cardiology and/or the emergency department for further evaluation. Further ECGs, cardiac biomarkers, cardiac imaging for such participants would be standard of care.

Assigning Subject Identification Numbers:

Upon consent, the subject will be randomly assigned a subject ID number. Subjects requiring concomitant vaccines along with JYNNEOS® will be randomly assigned to one of two groups (1:1 allocation) and that simple computer-generated randomization will be concealed to research staff. The link between subject ID numbers and their names and dates of consent will be maintained at the DHA-IHD research office in a locked filing cabinet within locked offices, and/or in secure, password-protected electronic files, only accessible to the research study team. The linkage document will be destroyed after completion of the final data analysis and IRB acknowledgment/approval of study closure.

Location and Personnel for Study Procedures:

Study procedures will be performed at Defense Health Agency-Immunization Healthcare Division sites or within their AOR by the DHA-IHD study team. (e.g., the Fort Bragg study team may travel to Camp Lejeune to enroll subjects once approved by Camp Lejeune Commanders/Leadership). All study assessments will be performed by members of the investigative team that are specifically designated to perform such activities according to site practices, local laws, and as designated on the appropriate study documents. The Principal Investigator, in collaboration with Associate Investigators and statistician, will be responsible for the interpretation of the statistical information.

Demographic and Medical Data:

Research study staff will collect initial demographics (including age, sex, ethnicity, race, etc.), past medical history, height, weight, and vital signs (such as heart rate, blood pressure, temperature, pulse oximetry and respiratory rate). Demographics will be collected via questionnaire on enrollment day only. Vitals and any updates in medical history will be collected on enrollment day and follow-up visits as well as with weekly email or text surveys (utilizing RedCap or other electronic data management systems as available). Subjects will be asked to provide the study team with information on any medications being used at the time of enrollment and throughout the duration of their participation in the research study. Subjects will be queried on a history of cardiac risk factors and cardiac and atopic disease and be consented for permission to review their medical records, specifically looking for past immunization history, past medical history of cardiac and atopic disease, cardiac risk factors (such as hypertension, smoking, hyperlipidemia, obesity, etc), allergy/atopic history, previous HIV testing, and other relevant medical information. HIV status is specifically queried due to the fact that prelicensure studies identified a higher risk of cardiac events in HIV-positive individuals compared to the general population. Further evaluating for a link between HIV status and the risk of myopericarditis is important in identifying possible risks in this population. The electronic medical records (such as AHLTA, MHS Genesis, CHCS, MEDPROS, ASIMS, MRRS, etc.) may be queried by the research team who may extract subject-specific data to the CRFs/eCRFs.

AQUA Allergy Questionnaire:

Based upon the research team's previous work (unpublished), atopy has been associated with a possible increased risk of vaccinia-induced myopericarditis. Furthermore, in a prelicensure study of JYNNEOSTM patients with atopic dermatitis, the manufacturer reported elevations of troponin in 14.6% of subjects which is significantly elevated above non-atopic patients. Given such, screening for atopy would provide additional information on whether this finding holds true. To this end, the study team will administer a validated instrument (AQUA: Allergy Questionnaire for Athletes) that has the ability to predict atopy with a fairly high degree of sensitivity (58.3%) and specificity (97.1%). [14] This questionnaire is preferable to any additional laboratory testing such as total and/or specific IgE and will allow us to avoid additional phlebotomy. The owner of the AQUA questionnaire has provided written permission to use this instrument for the study. The questionnaire will be administered at the initial visit. Additionally, medical history obtained on day of enrollment will ask about a history of hymenoptera hypersensitivity and drug allergies. Such data will be annotated in the CRF/eCRFs. See "other documents" for a copy of the AQUA questionnaire.

Blood Collection:

Subjects will undergo phlebotomy at each of the 5 visits over a 9-week (65 daytime period: once prior to vaccination (at visit 1) and on post-vaccination days 8-14 (visit 2), 28-34 (visit 3), 39-45 (visit 4) and 59-65 (visit 5). All specimens will be labeled with the subject's study identification number (no personal identifiers), type of specimen, date and time of collection, and visit number. Serum/plasma specimens will be processed appropriately and sent to the laboratory for testing. Currently, at the Fort Bragg site, specimen testing will be performed at the WAMC pathology laboratory. Batch processing of specimens for hsTnT may be coordinated with pathology as not to interfere with ongoing clinical care demands. Each stored tube will be tracked with a subject identification number linked database that includes sample type and location in freezer. All specimens will be handled and disposed of in accordance with federal regulations.

This study will use standard clinical blood profiles to determine clinical chemistry and blood markers associated with smallpox vaccination and myopericarditis. Up to ~140 mL (10 tablespoons) of whole blood will be obtained from all subjects via phlebotomy on the following schedule: ~28 mL (2 tablespoons) immediately prior to vaccination (visit 1), ~28 mL (2 tablespoons) between days 8-14 (visit 2), ~28 mL (2 tablespoons) 28-34 days following vaccination # 1 in the series but before vaccination #2 in the series (visit 3), ~28 mL (2 tablespoons) again at day 39-45 (visit 4), and a final draw of ~28 mL (2 tablespoons) at day 59-65 (visit 5).

The following laboratory studies will be conducted at the initial visit once enrolled and prior to vaccination to include standard hematological (CBC with differential) and clinical chemistry markers (Complete Metabolic Profile and Creatinine Phosphokinase) to ensure baseline healthy subjects as well as various myocardial injury markers to include high sensitivity Troponin I (hsTnI), high sensitivity Troponin T (hsTnT) and high sensitivity C-reactive protein (hsCRP). In addition, all follow-up visits will include additional laboratory studies which include the various myocardial injury markers mentioned above to include high sensitivity Troponin I (hsTnI), high sensitivity Troponin T (hsTnT) and high sensitivity C-reactive protein (hsCRP). Primary blood profile endpoints will include mean values of the markers at baseline and correlation between changes in biochemical immunization. Secondary blood profile endpoints will include association with clinical outcomes. Clinical outcomes will include, but not be limited to, referral for evaluation of cardiovascular disease within 30 days post immunization, as well as further analysis to assess possible covariates that may be observed in the initial data analysis.

The research team will conduct all studies using these specimens as research only. However, in the event of an abnormal value identified on baseline labs, the labs will be reviewed by a clinical provider on the research team and the results of the abnormal labs may be relayed to the patient as well as the suggested best course of action for further evaluation (such as scheduling an appointment with the PCM, urgent care or emergency department visit). Labs performed at the local MTF will be entered in CHCS under a research name and number specific to the subject ID and visit number. These lab results will not be reflected in the actual subject's electronic health record under their name, DoD ID, or Social Security number. Every effort will be made to protect confidentiality and no one other than the research team or the Principal Investigator will receive results of the test, with the exceptions noted above for abnormal values. Of note, interpretation of a hsTnT value at a single point in time can be difficult. The diagnostic importance is the change (delta) of the hsTroponin over time. To increase the validity of any significant changes in troponin the research team may batch process specimens so all testing from all 5 visits of an individual subject's specimens are run at the same time (same assay, same machine in same laboratory day) to decrease variability introduced by different assays, different calibrations, lab personnel handling, etc. Though doing so increases sensitivity of detecting significant changes, it also prohibits timely identification of subclinical myopericarditis in a subject. However, given troponin testing is not considered part of the standard of care following any smallpox vaccination and given the clinical significance of an elevated hsTroponin level post-immunization without any accompanying symptoms or ECG changes is not known, and given that the FDA did not require any additional observational studies looking for myocardial injury in JYNNEOSTM vaccinees the investigators feel the risk of such an approach is minimal. Subjects who report clinical symptoms and/or who have abnormal ECG readings would be referred to DHA-IHD clinical teams in consultation with cardiology for further evaluation and management of possible vaccinia-associated myopericarditis (standard of care).

Visit 1/baseline labs Certain laboratory tests will be performed at visit 1 only and will be processed in the local lab or reference labs. These baseline labs tests include a complete blood count (CBC) with differential, comprehensive metabolic profile (CMP), creatinine phosphokinase (CPK), and hsCRP. At the Fort Bragg site, these tests will be performed by WAMC Pathology via the agreement on their impact statement. The CBC and differential will be used to define the baseline lymphocyte count. The initial hematology profile and the CMP will also be utilized to help us understand the population health preimmunization (i.e., rule out underlying kidney, liver or metabolic disease that might alter some of the other biomarkers). Samples will be handled for rapid submission to the study site local medical treatment facility laboratory (CBC, CMP) and for local storage prior to batch processing (hsTnT, CPK and hsCRP) to avoid error due to degradation prior to testing. Batch processing will permit sample testing to be performed in tandem with the same assay allowing for more sensitive evaluations in changes of biomarkers. Also, based upon the WAMC pathology impact statement, the hsTnT labs will have to be coordinated as not to impact clinical care demands for this test. Of note, hsTnI is not readily available at the current time as it was just recently FDA-approved and this test is not available at any current MTF or common send-out labs such as LabCorp. Therefore, plasma for this lab will initially be stored in DHA-IHD freezers (location previously identified) with plans for future testing as described above after any formal coordination and agreements have been completed. A protocol modification will be submitted and approved before any hsTnI testing is conducted as part of this clinical study.

Follow-up visit labs; visits 2-5 Follow-up laboratory tests will be performed in the local or reference lab due to the investigatory nature of some of these biomarkers. (For the Fort Bragg site, these tests will be run at the WAMC laboratory). These tests include hsTnT, hsCRP and CPK. Plasma/serum assays for CPK and hsCRP are routine commercially available tests, with independent quality assurance provided both by the manufacturer and performed within any standard laboratory. High sensitivity TnI and hsTnT may be performed at the local MTF or sent to a reference lab depending on the current capabilities of the labs during the 4-5 year study period. Samples will be handled for rapid processing and local storage prior to batch processing (hsTnT, hsCRP and CPK) to avoid error due to degradation prior to testing. Batch processing will permit sample testing to be performed in tandem with the same assay allowing for more sensitive evaluations in changes of these biomarkers. Of note, hsTnI is not readily available at the current time as it was just recently FDA-approved and this test is not available at any current MTF or common send-out labs such as LabCorp. Therefore, serum for this lab with initially be stored in DHA-IHD freezers with plans for future testing as described above after any formal coordination and agreements have been completed. A protocol modification will be submitted and approved before any hsTnI testing is conducted as part of this clinical study.

Electrocardiogram (ECG) Subjects will undergo a 12-lead ECG at every visit. Standard 12-lead ECGs will be performed using certified local clinic-based equipment. The results will not be disclosed to the subject as this is a study-related procedure and not standard of care. A cardiologist will review all ECG tests but readings may not occur in real-time and may be batch read at a later date which could be weeks or months after the actual ECG was obtained. However, if a machine reading identifies a significant abnormality (such as arrhythmia, pericarditis, acute myocardial injury, etc.) the study team will notify a study investigator to review the machine-identified abnormality as soon as possible. The study investigator can provide further recommendations, such as seeking care from the primary care manager, emergency room, or the Defense Health Agency-Immunization Healthcare Division vaccine safety hub clinic. ECG tracings from all available visits may be reviewed in a single session to rectify inaccurate machine reads when appropriate, and to validate changes from baseline as one might expect with vaccinia-induced myopericarditis. ECGs showing changes consistent with pericarditis and/or myocarditis may undergo a second blinded review by a different cardiologist. Cardiologists interpreting the ECGs will be blinded to the allocation of group assignment for those subjects requiring concomitant vaccines.

Symptom Surveys All subjects will be given an electronic link to a survey via RedCap or other electronic method to complete between visits to better surveil for myopericarditis symptoms. (see "other documents" for a sample of the survey). This survey will be distributed via email or text at the subjects preference. This diary/survey tool will keep track of any symptoms that may occur during the duration of the subject's participation. This symptom survey will ask if the subject is experiencing headaches, chest, back, shoulder or abdominal pains or discomfort, fatigue, shortness of breath, etc. Additionally, the diary/survey may ask about other systemic symptoms such as rashes, fevers, chills, and local adverse events such as lymphadenopathy and large local reactions. The Defense and Veterans Pain Rating Scale (DVPRS) will be utilized by the subjects to rate the level of their pain on a scale of 1 to 10. Links to the surveys will be sent at various times between clinical visits. Specifically, surveys will be sent once between visit 1 and visit 2 (at approximately day 5-6) , twice between visit 2 and visit 3 (at approximately day 17-18 and again approximately day 24-25) , once between visit 3 and visit 4 (at approximately day 36-37), and twice between visit 4 and visit 5 (at approximately day 49-50 and again at day 56-57). hsTnT/hsTnI testing from stored specimens of WAMC Protocol #375283. This study also plans to conduct hsTnT testing on plasma from previously obtained specimens from one of the research team's sister studies. Specifically, Protocol #375283, "A Pilot Study: Smallpox/Influenza Vaccination and Myopericardial Injury/Inflammation." This protocol and its respective informed consent document allowed for storage of specimens for future vaccine research and specifically stated subjects would not be given any notice of future use of the stored specimens. Given it is unknown how the immunization process may impact hsTnT results, a control population with a different vaccine other than smallpox vaccine, would be an important parameter to help provide additional context to the investigators findings of this prospective study. To that end, the investigators plan to run hsTnT and possibly hsTnI testing (when readily available and all agreements are in place) on 282 specimens (141 pre-influenza immunization and 141 post- influenza immunization) obtained from this previous protocol which has remained open at WAMC. This protocol was last reviewed via a modification and approved on 25 SEP 2019. Aliquots of specimens are maintained in DHA-IHD -80ºC freezers. Specimens would be identified, and thawed only after coordination with the laboratory for hsTnT testing at a time that is determined to not impact WAMC clinical care. hsTnI testing would only be completed after a modification to this protocol and after all appropriate agreements are in place.

Cardiac Magnetic Resonance Imaging (CMR) As discussed above, the clinical significance of subclinical myopericarditis is not known. However, one would intuitively suspect that an elevated postimmunization hsTroponin above a known normal baseline preimmunization hsTroponin might indicate myocardial injury. To further evaluate if subclinical myopericarditis is associated with myocardial inflammation/injury the investigators plan to evaluate a small sample of subjects (no more than 20) who have asymptomatic hsTroponin elevations and determine if these troponin elevations correlate with actual myocardial injury as determined by late gadolinium enhancement on CMR. Current data suggests that CMR is now the non-invasive gold standard to help determine a diagnosis of myopericarditis. Identifying if the subclinical troponin elevations correlate with inflammation/injury of the myocardium in CMR would be extremely valuable. CMR is not readily available at WAMC and all current CMR for Fort Bragg patients are sent to Duke. The investigators are in initial discussions with Duke Cardiology to collaborate on this portion of the study. Agreements and coordination for such will be pursued as the study matures and a protocol modification will be submitted prior to conducting this portion of the study This portion of the study is currently planned only for the Core site (WAMC) and a maximum of 20 subjects with asymptomatic hsTroponin will be evaluated with CMR.

Follow-Up Visits Subjects will be contacted via phone, text, or email for reminders of upcoming visits. In addition, subjects will receive an email or text with a link to a brief health survey screening for any signs or symptoms of myopericarditis (such as shortness of breath, chest, shoulder, back or abdominal pain, etc.) as described previously. Subjects will be reminded to contact their medical provider should they experience the following signs and/or symptoms: Chest, back, shoulder, or upper abdominal pain, pressure or discomfort; Rapid or abnormal heart rhythm; Shortness of breath, at rest or during physical activity; Fluid retention with swelling of the participants legs, ankles and feet; Fatigue; Headache, body aches, joint pain, a sore throat or diarrhea.

In the unlikely event a subject is hospitalized for any reason during the study and the study team is made aware, attempts will be made to visit the patient in the hospital by one of the research team members to determine the cause of hospitalization, (and any need to report the hospitalization as an adverse event to the IRB/HRPO) as well as to assess for a possible vaccine-associated adverse event. Should the inpatient stay occur during a visit window, the subject will be asked if he or she desires to remain in the study and if so, the respective visit will be conducted to include associated phlebotomy in the subject's hospital room or other appropriate and private location.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military personnel within the range of 18-45 years of age without limitations to gender or ethnicity.
* Primary vaccinee (receiving smallpox vaccine for the first time) with a force health protection requirement for the smallpox vaccination
* Medical screening for immunization completed and potential participant found eligible for immunization (standard of care)

Exclusion Criteria:

* Known contraindication to replication deficient smallpox vaccination based on FDA-approved package insert for JYNNEOS™ vaccine.
* No indication for replication deficient smallpox vaccination based on FDA-approved package insert for JYNNEOS, ACIP or DoD guidelines
* Secondary smallpox vaccinee (patients who had previously received any smallpox vaccine).
* Age less than 18 years or age greater than 45 years.
* Inability to provide informed consent.
* Presence of a moderate or severe acute illness with or without a fever
* Pregnancy: We will rely on the subject for an assessment of her pregnancy status, based on answers in the routine adult immunization screening questionnaire. (Screening by history is the current standard of care.)
* Scheduled deployment, PCS or TDY that would interfere with the respective follow-up visits. (no planned deployment, TDY or PCS for 65 days after enrollment/visit 1).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 2350 Active duty military personnel age 18 to 45 years meeting the eligibility criteria and having a current force health protection requirement for the smallpox vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 2350 (Estimated)
Dates: Start 2029-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | Within 35 days following the 2-dose series of a novel, replication-deficient (JYNNEOS™) smallpox vaccine
  Determine the number of participants with myocarditis or pericarditis defined by abnormal laboratory biomarkers (hsTn) or abnormal ECG that may or may not be accompanied by subjective reports of chest, back, shoulder or upper abdominal pain or discomfort following receipt of the 2-dose series of a novel, replication-deficient (Jynneos™) smallpox vaccination in a group of adult primary smallpox vaccines.
Primary Outcome | Within 35 days following the 2-dose series of a novel, replication-deficient (JYNNEOS™) smallpox vaccine
  Determine the number of participants with myocarditis or pericarditis defined by abnormal laboratory biomarkers (hsTn) or abnormal ECG that may or may not be accompanied by subjective reports of chest, back, shoulder or upper abdominal pain or discomfort following receipt of the 2-dose series of a novel, replication-deficient (Jynneos™) smallpox vaccination with co-receipt of any other ACIP recommended vaccine in a group of adult primary smallpox vaccines.

SECONDARY OUTCOMES:
Secondary Objective | Within 35 days following the 2-dose series of a novel, replication-deficient (JYNNEOS™) smallpox vaccine
  Compare the difference in prospective incidence of symptomatic or asymptomatic myopericarditis when the first dose of Jynneos™ smallpox vaccination is administered concomitantly with other required vaccines versus when the first dose of Jynneos is administered in isolation from other required vaccines by at least 28 days.
Tertiary Objective | Within 35 days following the 2-dose series of a novel, replication-deficient (JYNNEOS™) smallpox vaccine
  Determine the number of participants with changes in hsCRP and/or CPK and compare to hsTn, abnormal ECG changes and subjective reports of chest, back, shoulder or upper abdominal pain or discomfort following receipt of the 2-dose series of a novel, replication-deficient (Jynneos™) smallpox vaccination in a group of adult primary smallpox vaccines.
Quaternary Objective | Within 35 days following the 2-dose series of a novel, replication-deficient (JYNNEOS™) smallpox vaccine
  Measure the presence or absence of any late gadolium enhancement, and ejection fraction on cardiac MRI among participants who demonstrate abnormal laboratory biomarkers (hsTn) or abnormal ECG in the absence of subjective reports of chest, back, shoulder or upper abdominal pain or discomfort following receipt of the 2-dose series of a novel, replication-deficient (Jynneos™) smallpox vaccination in a group of adult primary smallpox vaccines.

REFERENCES:
- [Background] Casey C, Vellozzi C, Mootrey GT, Chapman LE, McCauley M, Roper MH, Damon I, Swerdlow DL; Vaccinia Case Definition Development Working Group; Advisory Committee on Immunization Practices-Armed Forces Epidemiological Board Smallpox Vaccine Safety Working Group. Surveillance guidelines for smallpox vaccine (vaccinia) adverse reactions. MMWR Recomm Rep. 2006 Feb 3;55(RR-1):1-16. PMID 16456528
- [Background] Halsell JS, Riddle JR, Atwood JE, Gardner P, Shope R, Poland GA, Gray GC, Ostroff S, Eckart RE, Hospenthal DR, Gibson RL, Grabenstein JD, Arness MK, Tornberg DN; Department of Defense Smallpox Vaccination Clinical Evaluation Team. Myopericarditis following smallpox vaccination among vaccinia-naive US military personnel. JAMA. 2003 Jun 25;289(24):3283-9. doi: 10.1001/jama.289.24.3283. PMID 12824210
- [Background] Godreuil S, Delhaume O, Besset-Prat L, Blayac JP, Peyriere H, Bonnet P. [Acute haemorrhagic pericarditis following influenza vaccination]. Presse Med. 2003 Feb 15;32(6):258-9. French. PMID 12610454
- [Background] Boccara F, Benhaiem-Sigaux N, Cohen A. Acute myopericarditis after diphtheria, tetanus, and polio vaccination. Chest. 2001 Aug;120(2):671-2. doi: 10.1378/chest.120.2.671. PMID 11502677
- [Background] Peyriere H, Hillaire-Buys D, Pons M, Navarre C, Davy JM, Blayac JP. [Acute pericarditis after vaccination against hepatitis B: a rare effect to be known]. Rev Med Interne. 1997;18(8):675-6. doi: 10.1016/s0248-8663(97)82474-5. No abstract available. French. PMID 9365747
- [Background] Helle EP, Koskenvuo K, Heikkila J, Pikkarainen J, Weckstrom P. Myocardial complications of immunisations. Ann Clin Res. 1978 Oct;10(5):280-7. PMID 736507
- [Background] Cono J, Casey CG, Bell DM; Centers for Disease Control and Prevention. Smallpox vaccination and adverse reactions. Guidance for clinicians. MMWR Recomm Rep. 2003 Feb 21;52(RR-4):1-28. PMID 12617510
- [Background] de Meester A, Luwaert R, Chaudron JM. Symptomatic pericarditis after influenza vaccination: report of two cases. Chest. 2000 Jun;117(6):1803-5. doi: 10.1378/chest.117.6.1803. PMID 10858422
- [Background] Feldman AM, McNamara D. Myocarditis. N Engl J Med. 2000 Nov 9;343(19):1388-98. doi: 10.1056/NEJM200011093431908. No abstract available. PMID 11070105
- [Background] Engler RJ, Nelson MR, Collins LC Jr, Spooner C, Hemann BA, Gibbs BT, Atwood JE, Howard RS, Chang AS, Cruser DL, Gates DG, Vernalis MN, Lengkeek MS, McClenathan BM, Jaffe AS, Cooper LT, Black S, Carlson C, Wilson C, Davis RL. A prospective study of the incidence of myocarditis/pericarditis and new onset cardiac symptoms following smallpox and influenza vaccination. PLoS One. 2015 Mar 20;10(3):e0118283. doi: 10.1371/journal.pone.0118283. eCollection 2015. PMID 25793705
- [Background] Grabenstein JD, Winkenwerder W Jr. US military smallpox vaccination program experience. JAMA. 2003 Jun 25;289(24):3278-82. doi: 10.1001/jama.289.24.3278. PMID 12824209
- [Background] Bonini M, Braido F, Baiardini I, Del Giacco S, Gramiccioni C, Manara M, Tagliapietra G, Scardigno A, Sargentini V, Brozzi M, Rasi G, Bonini S. AQUA: Allergy Questionnaire for Athletes. Development and validation. Med Sci Sports Exerc. 2009 May;41(5):1034-41. doi: 10.1249/MSS.0b013e318193c663. PMID 19346984
- [Background] Silverberg JI. Atopic disease and cardiovascular risk factors in US children. J Allergy Clin Immunol. 2016 Mar;137(3):938-40.e1. doi: 10.1016/j.jaci.2015.09.012. Epub 2015 Dec 8. No abstract available. PMID 26679356
- [Background] Xu RY, Zhu XF, Yang Y, Ye P. High-sensitive cardiac troponin T. J Geriatr Cardiol. 2013 Mar;10(1):102-9. doi: 10.3969/j.issn.1671-5411.2013.01.015. PMID 23610580
- See also: JYNNEOS package insert — https://www.fda.gov/media/131078/download